CLINICAL TRIAL: NCT05624463
Title: Effect of Modified Endotracheal Intubation Protocol Combined With Early Oral Intake on Postoperative Recovery Quality in Thyroid and Parathyroid Surgery at a Tertiary Hospital in China: A 2x2 Factorial Randomized Controlled Trial Protocol
Brief Title: Effect of Modified Endotracheal Intubation Protocol Combined With Early Oral Intake on Postoperative Recovery Quality in Thyroid and Parathyroid Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: K-2501
Record Dates: First submitted 2022-11-13; First posted 2022-11-22 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Thyroid Tumor
Keywords: Thyroidectomy; Enhanced Recovery After Surgery; Quality of Recovery-15; Parathyroidectomy
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial：Participants who enroll in randomized controlled trials differ from one another in known and unknown ways that can influence study outcomes, and yet cannot be directly controlled. By randomly allocating participants among compared treatments, an randomized controlled trial enables statistical control over these influences. Provided it is designed well, conducted properly, and enrolls enough participants, an randomized controlled trial may achieve sufficient control over these confounding factors to deliver a useful comparison of the treatments studied.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The questionnaire collectors and outcomes assessor will not be informed of the group of patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Modified intubation protocol+early resumption of oral intake (Experimental): Participants receive modified intubation protocol and early resumption of oral intake.
  Interventions: Behavioral: Modified intubation protocol; Behavioral: Early resumption of oral intake
- Modified intubation protocol+delayed resumption of oral intake (Other): Participants receive modified intubation protocol and delayed resumption of oral intake.
  Interventions: Behavioral: Modified intubation protocol; Behavioral: Delayed resumption of oral intake
- Conventional intubation protocol+early resumption of oral intake (Other): Participants receive conventional intubation protocol and early resumption of oral intake.
  Interventions: Behavioral: Conventional intubation protocol; Behavioral: Early resumption of oral intake
- Conventional intubation protocol+delayed resumption of oral intake (Other): Participants receive conventional intubation protocol and delayed resumption of oral intake.
  Interventions: Behavioral: Conventional intubation protocol; Behavioral: Delayed resumption of oral intake

INTERVENTIONS:
Behavioral: Modified intubation protocol — 1. Turn on the electromyography (EMG) monitor and connect the EMG monitor to the patient as the patient is anesthetized; 2. View the vocal cords with video laryngoscope and intubate the patient with the EMG endotracheal tube; 3. Check the EMG monitor to confirm the correct contact between the electrodes and vocal cords; 4. Adjust the tube to achieve proper and stable contact between the electrodes and vocal cords; 5. Tape the EMG endotracheal tube at the midline and position the patient.
  Arms: Modified intubation protocol+delayed resumption of oral intake; Modified intubation protocol+early resumption of oral intake
Behavioral: Conventional intubation protocol — 1. Intubate the patient with the EMG endotracheal tube and note depth; 2. Position patient and verify the position via Glottic Exam or Respiratory Variation; 3. Fix tube position.
  Arms: Conventional intubation protocol+delayed resumption of oral intake; Conventional intubation protocol+early resumption of oral intake
Behavioral: Early resumption of oral intake — Patients will drink 30-50ml of normal temperature water after Steward scores ≥ 4 at PACU. If patients swallow successfully and have no significant discomfort symptoms, physicians will guide patients to resume drinking and eating gradually.
  Arms: Conventional intubation protocol+early resumption of oral intake; Modified intubation protocol+early resumption of oral intake
Behavioral: Delayed resumption of oral intake — Patients will resume drinking water 6h after the operation at ward. Before patients resume oral drinking, they will be provided 10ml/kg 5% glucose saline intravenously.
  Arms: Conventional intubation protocol+delayed resumption of oral intake; Modified intubation protocol+delayed resumption of oral intake

SUMMARY:
The purpose of this study is to assess the effect of modified endotracheal intubation procedure combined with early oral intake on postoperative recovery quality of patients, so as to further optimize the ERAS（enhanced recovery after surgery） program for thyroid or parathyroid surgery.

DETAILED DESCRIPTION:
After being informed about the study and potential risk, all patients giving written informed consent will undergo a screening-period to determine eligibility for study entry. Before operation, patients will be randomly assigned to conventional intubation process group or modified intubation process group before the operation. After the operation, patients will enter the PACU（post-anaesthesia care unit） for further observation. When the anesthesiologists and surgeons agree that patients have no early oral drinking high-risk factors, patients will be randomly assigned to early resumption of oral intake group or late resumption of oral intake group for further observation and evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* American Society of Anesthesiologists (ASA) physical status classification I-II
* Body mass index 18.5-29.9kg/m2
* First operation on operation day

Exclusion Criteria:

* Patients or family members cannot understand the conditions and objectives of this study
* Preoperative patients with acute pharyngitis, hoarseness, cough, dysphagia, and high risk of aspiration
* The surgeons or anesthesiologists point out that the patient is not suitable for early postoperative drinking (such as considering the injury of recurrent laryngeal nerve or lymphatic vessels during the operation)
* Patients who cannot be intubated under visual laryngoscope(such as difficult airway, loose incisors and so on)
* Exclusion criteria of Quality of Recovery-15* (*Quality of Recovery-15 exclusion criteria: 1. Unable to understand words and language; 2. Difficult to cooperate due to mental disorders; 3. History of alcohol or drug abuse; 4. Any serious pre-existing medical condition that can limit the objective evaluation after surgery; 5. Any life-threatening complications; 6. Emergency surgery)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-02-06 (Actual); Study Completion 2024-02-09 (Actual)

PRIMARY OUTCOMES:
Quality of Recovery-15 score on the first day after surgery | one day
  Using Quality of Recovery-15 questionnaire to evaluate the quality of perioperative recovery. Quality of Recovery-15 consists of 15 comprehensive questions, including physical comfort (5 items), psychological support (2 items), physical independence (2 items), emotional state (4 items), and pain (2 items), each item is scored with 0-10 points, 0 represents poor state, 10 represents good state, and the total score is the Quality of Recovery-15 score of the patient.

SECONDARY OUTCOMES:
Quality of Recovery-15 score on the day of discharge | one day
  Using Quality of Recovery-15 questionnaire to evaluate the quality of perioperative recovery. Quality of Recovery-15 consists of 15 comprehensive questions, including physical comfort (5 items), psychological support (2 items), physical independence (2 items), emotional state (4 items), and pain (2 items), each item is scored with 0-10 points, 0 represents poor state, 10 represents good state, and the total score is the Quality of Recovery-15 score of the patient.
Patient satisfaction | through patient discharge, an average of 2-3 days after surgery
  Patient satisfaction was assessed based on the postoperative numeric rating scale (NRS) scores, with 0 indicating extreme dissatisfaction and 10 indicating very satisfaction.
Postoperative pain | one day
  The patients were given self-evaluation before resuming oral intake and one day after the surgery. Pharyngeal pain and surgical incision pain were assesed by a visual analogue scale (VAS), with 0 indicating no pain and 10 indicating the worst pain.
Postoperative patient discomfort | one day
  The postoperative patient discomfort included the feeling of thirst and hunger. The patients were given self-evaluation before surgery and before resuming oral intake after surgery. The discomfort feelings were assesed by a visual analogue scale (VAS), with 0 indicating no discomfort and 10 indicating the worst discomfort.
Intubation time | one day
  Time from the end of pre-oxygenation to the completion of intubation and position setted.
Endotracheal tube readjustment rate | one day
  Rate of endotracheal tube readjustment caused by the lose or weakness of monitor signal during the surgery.
Postoperative nausea and vomiting | through patient discharge, an average of 2-3 days after surgery
  Researchers recorded the occurences and treatments of postoperative nausea and vomiting.
Gastrointestinal recovery time | through exhaustion after surgery, an average of 1-2 days after surgery
  The first postoperative exhaustion time recorded was considered as gastrointestinal recovery time.
Drainage volume | through removal of drainage tube, an average of 2 days after surgery
  Total drainage volume after operation.
Postoperative hospital stay length | through patient discharge, an average of 2-3 days after surgery
  Postoperative hospital stay length
Adverse event | through patient discharge, an average of 2-3 days after surgery
  The occurrence of adverse events such as severe choking, reintubation, postoperative bleeding.

CONTACTS AND LOCATIONS:
Overall Officials: Le Shen, PhD, Study Chair — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication are to be shared to other researchers.
Supporting Information: Study Protocol
Time Frame: Starting 6 months after publication, and ending 24 months after publication.
Access Criteria: Researchers may apply for IPD after data access proposal was approved by Research Ethics Committee of PUMCH. IPD can be used for meta-analysis of individual participant data. Data access proposal should be sent to pumchshenle@163.com, and IPD will be returned to the applicants.

REFERENCES:
- [Derived] Wu J, Zhang Y, Shen L. Modified versus conventional intubation and early versus delayed oral intake in thyroid surgery: a 2 x 2 factorial randomized controlled trial. Perioper Med (Lond). 2025 Oct 9;14(1):106. doi: 10.1186/s13741-025-00594-w. PMID 41068829
- [Derived] Wu J, Zhang Y, Shen L. Effect of modified endotracheal intubation protocol combined with early oral intake on postoperative recovery quality in thyroid and parathyroid surgery at a tertiary hospital in China: a 2x2 factorial randomised controlled trial protocol. BMJ Open. 2024 Jan 18;14(1):e075999. doi: 10.1136/bmjopen-2023-075999. PMID 38238052